CLINICAL TRIAL: NCT01474148
Title: A Neuroprosthesis for Seated Posture and Balance
Acronym: Trunk Protocol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1204-R; IRB#07101-H36 (Other: Case Western Reserve University)
Record Dates: First submitted 2011-11-08; First posted 2011-11-18 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injury; Paralysis; Tetraplegia; Paraplegia
Keywords: paraplegia; tetraplegia; Spinal cord injured; FES
MeSH Terms: conditions — Spinal Cord Injuries; Paralysis; Quadriplegia; Paraplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Neuroprosthesis (Experimental): Volunteers are evaluated for appropriateness for inclusion in the study on an intent-to-treat basis. Qualifying candidates all receive the implanted neuroprosthesis and participate in post-operative training and follow-up procedures.
  Interventions: Device: IRS-8 (8-Channel implanted stimulator-telemeter)

INTERVENTIONS:
Device: IRS-8 (8-Channel implanted stimulator-telemeter) — Surgical implantation of the 8-channel neuroprosthesis
  Other Names: Implanted Neuroprosthesis for Seated Posture and Balance, Trunk implanted electrical stimulation system, Implanted trunk control neuroprosthesis, Implanted FNS

SUMMARY:
The purpose of this study is to evaluate a surgically implanted functional electrical stimulation (FES) system to facilitate stability of the trunk and hips. FES involves applying small electric currents to the nerves, which cause the muscles to contract. This study evaluates how stabilizing and stiffening the trunk with FES can change the way spinal cord injured volunteers sit, breathe, reach, push a wheelchair, or roll in bed.

DETAILED DESCRIPTION:
In a single surgical procedure electrodes will be inserted into muscles of the trunk and hip musculature. The electrode leads are connected to a stimulator/telemeter located in the abdomen. After a typical post-operative period of two to five days, neuroprosthesis recipients will be discharged to home for two to six weeks of restricted activity to promote healing of all surgical incisions. After a period of exercise and training, functional use of the neuroprosthesis will begin. Laboratory assessments of strength, balance, and functional abilities with and without the system, as well as the technical performance of the implanted components will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* C4-T12
* ASIA Scale A through C
* Time post injury greater than 6 months
* Innervated and excitable trunk and pelvis musculature
* Absence of acute or chronic psychological problems or chemical dependency
* Range of motion within normal limits
* Controlled spasticity and absence of hip flexion and adduction spasm
* Height and weight within normal limits
* No history of balance problems or spontaneous falls
* No history of spontaneous fracture or evidence low bone density
* No acute orthopaedic problems
* No acute medical complications
* Adequate social support and stability
* Able to speak and read English

Exclusion Criteria:

* Pregnancy
* Non-English speaking

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-11-30 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Effect of Trunk stimulation on control seated posture, respiration, seated interface pressures, reach ability, seated stability & personal mobility. | up to 36 months
  Experiments involving the effects of trunk stimulation on postural alignment; trunk stability and posture on respiration, postural variation on seated interface pressures; effects of trunk stimulation on reaching ability; effects of trunk stimulation on seated stability, and personal mobility.

SECONDARY OUTCOMES:
Design a simple position controller | Up to 36 months
  The position controller will be developed to keep the trunk posture at a neutral seated position while allowing movement to lean forward, backward, or side-to-side. Testing will be carried out with an automated pull system applied to the trunk which pulls the body in various ways (side-to-side, forward, backward)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Triolo, PhD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Triolo RJ, Boggs L, Miller ME, Nemunaitis G, Nagy J, Bailey SN. Implanted electrical stimulation of the trunk for seated postural stability and function after cervical spinal cord injury: a single case study. Arch Phys Med Rehabil. 2009 Feb;90(2):340-7. doi: 10.1016/j.apmr.2008.07.029. PMID 19236990
- [Background] Bogie KM, Triolo RJ. Effects of regular use of neuromuscular electrical stimulation on tissue health. J Rehabil Res Dev. 2003 Nov-Dec;40(6):469-75. doi: 10.1682/jrrd.2003.11.0469. PMID 15077659
- [Derived] Foglyano KM, Lombardo LM, Schnellenberger JR, Triolo RJ. Sudden stop detection and automatic seating support with neural stimulation during manual wheelchair propulsion. J Spinal Cord Med. 2022 Mar;45(2):204-213. doi: 10.1080/10790268.2020.1800278. Epub 2020 Aug 14. PMID 32795162
- [Derived] Armstrong KL, Lombardo LM, Foglyano KM, Audu ML, Triolo RJ. Automatic application of neural stimulation during wheelchair propulsion after SCI enhances recovery of upright sitting from destabilizing events. J Neuroeng Rehabil. 2018 Mar 12;15(1):17. doi: 10.1186/s12984-018-0362-2. PMID 29530053
- [Derived] Triolo RJ, Bailey SN, Foglyano KM, Kobetic R, Lombardo LM, Miller ME, Pinault G. Long-Term Performance and User Satisfaction With Implanted Neuroprostheses for Upright Mobility After Paraplegia: 2- to 14-Year Follow-Up. Arch Phys Med Rehabil. 2018 Feb;99(2):289-298. doi: 10.1016/j.apmr.2017.08.470. Epub 2017 Sep 9. PMID 28899825
- [Derived] Wu GA, Lombardo L, Triolo RJ, Bogie KM. The effects of combined trunk and gluteal neuromuscular electrical stimulation on posture and tissue health in spinal cord injury. PM R. 2013 Aug;5(8):688-96. doi: 10.1016/j.pmrj.2013.03.025. Epub 2013 Mar 28. PMID 23542776
- [Derived] Triolo RJ, Bailey SN, Miller ME, Lombardo LM, Audu ML. Effects of stimulating hip and trunk muscles on seated stability, posture, and reach after spinal cord injury. Arch Phys Med Rehabil. 2013 Sep;94(9):1766-75. doi: 10.1016/j.apmr.2013.02.023. Epub 2013 Mar 13. PMID 23500182
- See also: Cleveland FES center website — http://fescenter.org